CLINICAL TRIAL: NCT04452877
Title: An Open-Label, Single-arm Study to Evaluate the Safety and Efficacy of Dabrafenib in Combination With Trametinib in Chinese Patients With BRAF V600E Mutation-Positive Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of Dabrafenib in Combination With Trametinib in Chinese Patients With BRAF V600E Mutant Metastatic NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDRB436ECN01
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Metastatic Non-Small Cell Lung Cancer; NSCLC; Chinese patients; dabrafenib; trametinib; BRAF V600E; treatment naive; pre-treated
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dabrafenib in combination with trametinib (Experimental): Dabrafenib 150 mg twice daily, trametinib 2 mg once daily
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Dabrafenib will be provided by the sponsor to the investigative site or supplied locally as commercially available. Dabrafenib will be administered orally twice daily (150 mg BID) for Days 1-21 of a 21-day cycle.
  Other Names: DRB436
Drug: Trametinib — Trametinib will be provided by the sponsor to the investigative site or supplied locally as commercially available. Trametinib will be administered orally once daily (2 mg QD) for Days 1-21 of a 21-day cycle
  Other Names: TMT212

SUMMARY:
This was a single-arm, open label, multicenter phase II, study of dabrafenib in combination with trametinib in Chinese participants with BRAF V600E mutation positive, stage IV NSCLC (American joint committee on cancer staging 8th edition). Approximately 40 Chinese adults were to be enrolled in this study. Participants were to be treated with dabrafenib in combination with trametinib until disease progression, start of a new anti-neoplastic therapy, unacceptable toxicity, pregnancy, withdrawal of consent, lost to follow-up, physician's decision, death, or if study be terminated by the sponsor. The general study design was discussed and agreed with China National Medical Products Administration and was based on a similar design used in the global pivotal phase II study (Study 113928 / NCT01336634).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of Stage IV NSCLC (according to AJCC 8th edition) that is BRAF V600E mutation-positive by local test result from a qualified assay (NMPA and/or MOH-approved)
* Previously treated or untreated for metastatic NSCLC:

  1. Participants previously treated should have received no more than 3 prior systemic therapies for metastatic disease, with at least one prior platinum based chemotherapy, and should have documented disease progression on a prior treatment regimen (i.e. RECIST 1.1)
  2. Participants who have received prior therapy with checkpoint inhibitor therapy (i.e. anti-PD-1/PD-L1) must have had objective evidence of disease progression (i.e. RECIST v1.1) while on or after this therapy prior to enrollment.
  3. Participants with EGFR or ALK mutation who have previously received therapy with EGFR or ALK inhibitor(s) respectively are eligible
* Measurable disease per RECIST v1.1
* Anticipated life expectancy of at least 3 months
* ECOG performance status ≤ 2.
* Adequate bone marrow and organ function as defined by the following laboratory values without continuous supportive treatment (such as blood transfusion, coagulation factors and/or platelet infusion, or red/white blood cell growth factor administration) as assessed by local laboratory for eligibility: Hemoglobin ≥ 9 g/dL; Absolute neutrophil count ≥ 1.5 × 109/L; Platelets ≥ 100 × 109/L; PT/INR and PTT ≤ 1.5 x ULN; Serum creatinine < 1.5 mg/dL; Total bilirubin ≤ 1.5 × ULN (upper limit of normal) except for participants with Gilbert's syndrome who may only be included if the total bilirubin is ≤ 3.0 × ULN or direct bilirubin ≤ 1.5 × ULN; AST and ALT ≤ 2.5 × ULN, except for participant with liver metastasis, who may only be included if AST/ALT ≤ 5.0 × ULN Albumin ≥ 2.5 g/dL
* Left ventricular ejection fraction (LVEF) ≥ lower limit of institutional normal (LLN) as assessed by ECHO or MUGA scan

Exclusion Criteria:

* Participants with brain or leptomeningeal metastases are excluded if their these metastases are: symptomatic or treated but not clinically and radiographically stable 3 weeks after local therapy or asymptomatic and untreated but >1 cm in the longest dimension
* Previous treatment with a BRAF inhibitor or a MEK inhibitor
* All prior anti-cancer treatment-related toxicities must be Grade 2 or less according to the Common Terminology Criteria for Adverse Events version 4 (CTCAE version 4.03; NCI, 2009) at the time of enrollment
* Prior anti-cancer treatment within the last 2 weeks, and prior treatment with immune checkpoint inhibitors within 4 weeks preceding the first dose of the study treatment.
* Current use of a prohibited medication
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO).
* Participants with known history for testing positive for Human Immunodeficiency Virus (HIV)
* History of another malignancy <3 years prior to starting study treatment or any malignancy with confirmed activating RAS-mutation.
* Cardiac or cardiac repolarization abnormality
* A history or current evidence/risk of retinal vein occlusion (RVO) or serous retinopathy
* History or current interstitial lung disease or non-infectious pneumonitis
* Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that, in the opinion of the investigator, could interfere with the participant's safety, obtaining informed consent, or compliance with study procedures
* Pregnant or nursing (lactating) women.
* Sexually active males (including those that have had a vasectomy) must use a condom during intercourse and should not father a child during this period. The amount of time a patient must use a condom for 16 weeks post treatment discontinuation
* Participants with active Hepatitis B infection (HbsAg positive)
* Participants with positive test for hepatitis C ribonucleic acid (HCV RNA)
* Concurrent participation in other clinical trials using experimental therapies

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- China (7):
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Result] Fan Y, Zhou J, Zhao Y, Yu Y, Yang N, Li J, Wang J, Zhao J, Wang Z, Chen J, Zhu T, Li H, Passos VQ, Bury-Maynard D, Zhang L. Efficacy, safety, and quality of life of dabrafenib plus trametinib treatment in Chinese patients with BRAF V600E mutation-positive metastatic non-small cell lung cancer. Transl Lung Cancer Res. 2024 Dec 31;13(12):3382-3391. doi: 10.21037/tlcr-24-494. Epub 2024 Dec 27. PMID 39830765
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2996

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 7 centers in China.
Period: Overall Study
Arm/Group | Dabrafenib in Combination With Trametinib
Started (All enrolled participants were included in the Full Analysis Set (FAS)) | 40
Pharmacokinetic Analysis Set (PAS) (Participants in the FAS for whom a PK sample was obtained and analyzed) | 38
Completed | 9
Not Completed | 31
Not completed — Adverse Event | 5
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 4
Not completed — Progressive Disease | 18
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Dabrafenib in Combination With Trametinib
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.1 (7.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 40

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR), Central Independent Review Assessed by RECIST v1.1
Description: Overall Response Rate (ORR) was defined as the proportion of participants with best overall response (BOR) of complete response (CR) or partial response (PR), as per central independent review assessment and according to RECIST 1.1.
Time Frame: From baseline until disease progression, death, lost to follow-up or withdrawal of consent, whichever occurs first, assessed up to approximately 50 months from treatment initiation
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage (%) of responders
Arm/Group | Dabrafenib in Combination With Trametinib
Number analyzed (Participants) | 40
Percentage (%) of responders | 75 [58.8 to 87.3]

2. Secondary Outcome: Overall Response Rate (ORR), Investigator Assessed by RECIST v1.1
Description: Overall Response Rate (ORR) was defined as the proportion of participants with best overall response (BOR) of complete response (CR) or partial response (PR) by Investigator assessment as per RECIST 1.1 criteria.
Time Frame: as for outcome 1
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage (%) of responders
Arm/Group | Dabrafenib in Combination With Trametinib
Number analyzed (Participants) | 40
Percentage (%) of responders | 77.5 [61.5 to 89.2]

3. Secondary Outcome: Progression Free Survival (PFS), Investigator Assessed by RECIST v1.1
Description: Progression Free Survival (PFS) was defined as the time from the date of first dose to the date of the first documented progression or death due to any cause. PFS was assessed via local review according to RECIST 1.1. PFS was censored if no PFS event was observed before the first to occur between: (i) the analysis cut-off date, and (ii) the date when a new anti-neoplastic therapy is started. The censoring date was the date of the last adequate tumor assessment prior to cut-off/start of new anti-neoplastic therapy.
Time Frame: From baseline until disease progression or death due to any cause, whichever occurs first, assessed up to approximately 50 months from treatment initiation
Population: Full Analysis Set (FAS)
Measure: Median (Full Range); unit: Months
Arm/Group | Dabrafenib in Combination With Trametinib
Number analyzed (Participants) | 40
Months | 13.9 [10.2 to 28.3]

4. Secondary Outcome: Duration of Response (DoR), Investigator Assessed by RECIST v1.1
Description: Duration of Response (DoR) only applies to participants whose Best Overall Response (BOR) was complete response (CR) or partial response (PR) according to RECIST 1.1 based on tumor response data per local review. The start date is the date of first documented response of CR or PR (i.e. the start date of response, not the date when response was confirmed), and the end date is defined as the date of the first documented progression or death due to any cause. Participants continuing without progression or death were censored at the date of their last adequate tumor assessment.
Time Frame: From first documented response until first documented progression or death due to any cause, whichever occurs first, assessed up to approximately 50 months from treatment initiation
Population: Full Analysis Set (FAS) - Subset of participants per local review with confirmed Best Overall Response (BOR) of complete response (CR) or partial response (PR)
Measure: Median (Full Range); unit: Months
Arm/Group | Dabrafenib in Combination With Trametinib
Number analyzed (Participants) | 31
Months | 14.9 [9.2 to 29.7]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time from date of first dose to date of death due to any cause. If a participant was not known to have died, then OS was censored at the latest date the participant was known to be alive (on or before the cut-off date).
Time Frame: From baseline until death due to any cause, assessed up to approximately 50 months from treatment initiation
Population: Full Analysis Set (FAS)
Measure: Median (Full Range); unit: Months
Arm/Group | Dabrafenib in Combination With Trametinib
Number analyzed (Participants) | 40
Months | 25.3 [16.2 to NA] — NA: Not estimable due to number of events censored

6. Secondary Outcome: Trough Concentration of Dabrafenib
Description: Plasma concentration of dabrafenib were calculated by visit/sampling time point and summarized using descriptive statistics.
Time Frame: Pre-dose sample at visits week 3, 6 and 12
Population: Pharmacokinetic Analysis Set (PAS) - Participants with corresponding evaluable PK parameters
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabrafenib in Combination With Trametinib
Number analyzed (Participants) | 38
ng/mL
  Week 3 (0 hours pre-dose): number analyzed (Participants) | 30
  Week 3 (0 hours pre-dose) | 74.4 (74.9)
  Week 6 (0 hours pre-dose): number analyzed (Participants) | 30
  Week 6 (0 hours pre-dose) | 91.5 (109.7)
  Week 12 (0 hours pre-dose): number analyzed (Participants) | 25
  Week 12 (0 hours pre-dose) | 93.9 (212.0)

7. Secondary Outcome: Trough Concentration of Dabrafenib Metabolites (Hydroxy-dabrafenib, and Desmethyl-dabrafenib)
Description: Plasma concentration of dabrafenib metabolites (hydroxy-dabrafenib, and desmethyl-dabrafenib) were calculated by visit/sampling time point and summarized using descriptive statistics.
Time Frame: Pre-dose sample at visits week 3, 6 and 12
Population: Pharmacokinetic Analysis Set (PAS) - Participants with corresponding evaluable PK parameters
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabrafenib in Combination With Trametinib
Number analyzed (Participants) | 38
ng/mL
  hydroxy-dabrafenib @ Week 3 (0 hours pre-dose): number analyzed (Participants) | 30
  hydroxy-dabrafenib @ Week 3 (0 hours pre-dose) | 81.9 (64.7)
  hydroxy-dabrafenib @ Week 6 (0 hours pre-dose): number analyzed (Participants) | 30
  hydroxy-dabrafenib @ Week 6 (0 hours pre-dose) | 93.8 (83.3)
  hydroxy-dabrafenib @ Week 12 (0 hours pre-dose): number analyzed (Participants) | 25
  hydroxy-dabrafenib @ Week 12 (0 hours pre-dose) | 100 (135.6)
  desmethyl-dabrafenib @ Week 3 (0 hours pre-dose): number analyzed (Participants) | 30
  desmethyl-dabrafenib @ Week 3 (0 hours pre-dose) | 510 (81.4)
  desmethyl-dabrafenib @ Week 6 (0 hours pre-dose): number analyzed (Participants) | 30
  desmethyl-dabrafenib @ Week 6 (0 hours pre-dose) | 468 (69.2)
  desmethyl-dabrafenib @ Week 12 (0 hours pre-dose): number analyzed (Participants) | 25
  desmethyl-dabrafenib @ Week 12 (0 hours pre-dose) | 430 (100.9)

8. Secondary Outcome: Trough Concentration of Trametinib
Description: Plasma concentration of trametinib were calculated by visit/sampling time point and summarized using descriptive statistics.
Time Frame: Pre-dose sample at visits week 3, 6 and 12
Population: Pharmacokinetic Analysis Set (PAS) - Participants with corresponding evaluable PK parameters
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabrafenib in Combination With Trametinib
Number analyzed (Participants) | 38
ng/mL
  Week 3 (0 hours pre-dose): number analyzed (Participants) | 32
  Week 3 (0 hours pre-dose) | 12.7 (35.0)
  Week 6 (0 hours pre-dose): number analyzed (Participants) | 31
  Week 6 (0 hours pre-dose) | 13.0 (29.5)
  Week 12 (0 hours pre-dose): number analyzed (Participants) | 26
  Week 12 (0 hours pre-dose) | 11.7 (37.0)

9. Secondary Outcome: Mean Change From Baseline in the European Quality of Life (EuroQol)- 5 Dimensions, 5 Level Questionnaire (EQ-5D-5L)
Description: The EQ-5D-5L is a standardized tool for measuring health-related quality of life (HRQoL). The instrument includes a descriptive system and a visual analogue scale. The descriptive system covers five dimensions (Mobility, Self-care, Usual activities, Pain/discomfort, Anxiety/depression), each with five severity levels ranging from 0 (no problems) to 5 (extreme problems) resulting in a 5-digit health code. In China, a country-specific value set is used to convert the five-digit health state into a utility score, ranging from <0 (worse than death) to 1.0 (perfect health). A positive change from baseline indicates improvement; a negative change indicates deterioration. The Visual Analog Scale (VAS) is a 0-100 self-rated health scale, where 0 is the worst and 100 the best imaginable health. A positive change reflects perceived improvement.
Time Frame: Baseline (BL), Week 12, End of Treatment (up to approximately 50 months after treatment initiation)
Population: Full Analysis Set (FAS) - Subset of participants with evaluable data at the pre-specified time points
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Dabrafenib in Combination With Trametinib
Number analyzed (Participants) | 33
Score on a Scale
  Mobility - Change from BL @ Week 12 | -0.09 (0.631)
  Mobility - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 18
  Mobility - Change from BL @ End of Treatment (EOT) Disposition | 0.06 (0.725)
  Self-Care - Change from BL @ Week 12 | 0.33 (0.174)
  Self-Care - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 18
  Self-Care - Change from BL @ End of Treatment (EOT) Disposition | 0.11 (0.323)
  Usual Activities - Change from BL @ Week 12 | 0.00 (0.433)
  Usual Activities - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 18
  Usual Activities - Change from BL @ End of Treatment (EOT) Disposition | 0.17 (0.383)
  Pain/Discomfort - Change from BL @ Week 12 | -0.33 (0.816)
  Pain/Discomfort - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 18
  Pain/Discomfort - Change from BL @ End of Treatment (EOT) Disposition | -0.17 (0.618)
  Anxiety/Depression - Change from BL @ Week 12 | -0.03 (0.467)
  Anxiety/Depression - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 18
  Anxiety/Depression - Change from BL @ End of Treatment (EOT) Disposition | 0.11 (0.583)
  Visual Analog Scale (VAS) - Change from BL @ Week 12 | 1.09 (8.611)
  Visual Analog Scale (VAS) - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 18
  Visual Analog Scale (VAS) - Change from BL @ End of Treatment (EOT) Disposition | -1.33 (10.000)

10. Secondary Outcome: Mean Change From Baseline in the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) Global Health Status/Quality of Life (GHS/QoL) Scale
Description: The EORTC QLQ-C30 is a 30-item questionnaire that patients complete, consisting of both multi-item scales and single-item measures. It includes five functional scales, three symptom scales, six single items, and a Global Health Status/Quality of Life (GHS/QoL) scale. The GHS/QoL scale has seven possible response scores ranging from 1 (very poor) to 7 (excellent), which are averaged and transformed to a 0-100 scale. A higher score on this scale indicates a better quality of life. The change from baseline in GHS/QoL scores is calculated. A positive change from baseline indicated improvement in the patient's quality of life.
Time Frame: Baseline (BL), Week 12, End of Treatment (up to approximately 50 months after treatment initiation)
Population: Full Analysis Set (FAS) - Subset of participants with evaluable data at the pre-specified time points
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Dabrafenib in Combination With Trametinib
Number analyzed (Participants) | 33
Score on a Scale
  Global Health Status - Change from BL @ Week 12 | 0.18 (0.882)
  Global Health Status - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 18
  Global Health Status - Change from BL @ End of Treatment (EOT) Disposition | -0.06 (0.938)
  Quality of Life - Change from BL @ Week 12 | 0.06 (0.747)
  Quality of Life - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 18
  Quality of Life - Change from BL @ End of Treatment (EOT) Disposition | -0.28 (0.669)

11. Secondary Outcome: Mean Change From Baseline in the European Organization for Research and Treatment of Cancer Lung Cancer Specific Module (EORTC QLQ-LC13)
Description: The EORTC QLQ-LC13 is a lung cancer-specific module designed to supplement the EORTC QLQ-C30 core questionnaire. It focuses on symptoms and side effects particularly relevant to lung cancer patients, including: Cough, Dyspnea (Shortness of breath), Hemoptysis (Coughing up blood), Sore Mouth/Tongue, Dysphagia (Trouble swallowing), Peripheral neuropathy (Tingling Hands/Feet), Alopecia (Hair Loss) and Pain in chest, arm, shoulder, or other areas and an additional dimension (Q13A: "How much did the pain medication help") if Q13: "did you take any medicine for pain" is answered "yes". Each item is scored on a 1 to 4 Likert scale (1 = "Not at all", 4 = "Very much") and then linearly transformed to a 0-100 scale. Improvements in QoL are indicated by decreased scores for the 13 main dimensions and an increased score for question 13A.
Time Frame: Baseline (BL), Week 12, End of Treatment (up to approximately 50 months after treatment initiation)
Population: Full Analysis Set (FAS) - Subset of participants with evaluable data at the pre-specified time points
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Dabrafenib in Combination With Trametinib
Number analyzed (Participants) | 33
Score on a Scale
  Cough - Change from BL @ Week 12 | -0.52 (0.712)
  Cough - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 17
  Cough - Change from BL @ End of Treatment (EOT) Disposition | -0.65 (0.606)
  Cough up blood - Change from BL @ Week 12 | -0.12 (0.331)
  Cough up blood - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 17
  Cough up blood - Change from BL @ End of Treatment (EOT) Disposition | 0.00 (0.000)
  Shortness of breath when resting - Change from BL @ Week 12 | -0.03 (0.394)
  Shortness of breath when resting - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 17
  Shortness of breath when resting - Change from BL @ End of Treatment (EOT) Disposition | 0.12 (0.332)
  Shortness of breath when walking - Change from BL @ Week 12 | -0.12 (0.650)
  Shortness of breath when walking - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 17
  Shortness of breath when walking - Change from BL @ End of Treatment (EOT) Disposition | 0.00 (0.791)
  Shortness of breath when climbing stairs - Change from BL @ Week 12 | -0.09 (0.805)
  Shortness of breath when climbing stairs - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 17
  Shortness of breath when climbing stairs - Change from BL @ End of Treatment (EOT) Disposition | -0.18 (0.809)
  Sore Mouth/Tongue - Change from BL @ Week 12 | 0.03 (0.305)
  Sore Mouth/Tongue - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 17
  Sore Mouth/Tongue - Change from BL @ End of Treatment (EOT) Disposition | 0.06 (0.243)
  Trouble swallowing - Change from BL @ Week 12 | -0.03 (0.305)
  Trouble swallowing - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 17
  Trouble swallowing - Change from BL @ End of Treatment (EOT) Disposition | -0.06 (0.429)
  Tingling Hands/Feet - Change from BL @ Week 12 | 0.06 (0.348)
  Tingling Hands/Feet - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 17
  Tingling Hands/Feet - Change from BL @ End of Treatment (EOT) Disposition | 0.29 (0.686)
  Hair Loss - Change from BL @ Week 12 | -0.03 (0.394)
  Hair Loss - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 17
  Hair Loss - Change from BL @ End of Treatment (EOT) Disposition | -0.06 (0.556)
  Pain in chest - Change from BL @ Week 12 | -0.15 (0.508)
  Pain in chest - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 17
  Pain in chest - Change from BL @ End of Treatment (EOT) Disposition | -0.06 (0.429)
  Pain in Arm/Shoulder - Change from BL @ Week 12 | -0.18 (0.528)
  Pain in Arm/Shoulder - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 17
  Pain in Arm/Shoulder - Change from BL @ End of Treatment (EOT) Disposition | -0.06 (0.659)
  Pain in Other Body Areas - Change from BL @ Week 12 | -0.30 (0.585)
  Pain in Other Body Areas - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 17
  Pain in Other Body Areas - Change from BL @ End of Treatment (EOT) Disposition | -0.35 (0.493)
  Any medicine for pain? - Change from BL @ Week 12 | -0.21 (0.415)
  Any medicine for pain? - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 17
  Any medicine for pain? - Change from BL @ End of Treatment (EOT) Disposition | -0.06 (0.429)
  Pain Medication Helpful? - Change from BL @ Week 12: number analyzed (Participants) | 3
  Pain Medication Helpful? - Change from BL @ Week 12 | 0.67 (0.577)
  Pain Medication Helpful? - Change from BL @ End of Treatment (EOT) Disposition: number analyzed (Participants) | 2
  Pain Medication Helpful? - Change from BL @ End of Treatment (EOT) Disposition | 0.50 (0.707)

12. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a participant or clinical investigation participant after providing written informed consent for participation in the study. Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product.
  Treatment Emergent Adverse Events (TEAEs) in this study are events that started after the first dose of study treatment and until 30 days after last dose.
Time Frame: From baseline until end of study, assessed up to approximately 50 months
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib in Combination With Trametinib
Number analyzed (Participants) | 40
Participants
  Adverse Events (AEs) | 39
  Treatment related AEs | 37
  AEs with grade >= 3 | 27
  Treatment related AEs with grade >= 3 | 18
  Serious Adverse Events (SAEs) | 20
  Treatment related SAEs | 11
  Fatal SAEs | 1
  Treatment related Fatal SAEs | 0
  Adverse Events (AEs) leading to discontinuation | 7
  Treatment related AEs leading to discontinuation | 5
  AEs leading to dose adjustment/interruption | 30
  AEs requiring additional therapy | 38

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from first dose of study medication until the last dose plus 30 days safety follow-up, assessed up to approximately 50 months. Deaths were recorded from study start date until end of post-treatment follow-up (end of study), assessed up to approximately 50 months. On-treatment period (up to 30 days after last dose) and post-treatment follow-up phase (thereafter) are reported separately.
Groups:
- Dabrafenib in Combination With Trametinib (On-treatment Period): Dabrafenib in combination with trametinib (On-treatment period): Events up to 30 days post-treatment
- Dabrafenib in Combination With Trametinib (Post-treatment Follow-up Phase): Dabrafenib in combination with trametinib (Post-treatment follow-up phase): Events in the post-treatment follow-up phase
Arm/Group | Dabrafenib in Combination With Trametinib (On-treatment Period) | Dabrafenib in Combination With Trametinib (Post-treatment Follow-up Phase)
All-Cause Mortality (participants affected / at risk) | 6/40 | 12/16
Serious Adverse Events (participants affected / at risk) | 20/40 | 1/16
Other Adverse Events (participants affected / at risk) | 39/40 | 1/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabrafenib in Combination With Trametinib (On-treatment Period) (N=40) | Dabrafenib in Combination With Trametinib (Post-treatment Follow-up Phase) (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Malaise (General disorders and administration site conditions) | 1 | 0
Pyrexia (General disorders and administration site conditions) | 5 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 0
Sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4.9999% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabrafenib in Combination With Trametinib (On-treatment Period) (N=40) | Dabrafenib in Combination With Trametinib (Post-treatment Follow-up Phase) (N=16)
Anaemia (Blood and lymphatic system disorders) | 21 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 3 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Ventricular extrasystoles (Cardiac disorders) | 3 | 0
Cataract (Eye disorders) | 4 | 0
Dry eye (Eye disorders) | 2 | 0
Optic disc haemorrhage (Eye disorders) | 2 | 0
Visual field defect (Eye disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Flatulence (Gastrointestinal disorders) | 3 | 0
Mouth ulceration (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 5 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Chest discomfort (General disorders and administration site conditions) | 2 | 0
Chest pain (General disorders and administration site conditions) | 2 | 0
Chills (General disorders and administration site conditions) | 2 | 0
Fatigue (General disorders and administration site conditions) | 4 | 0
Influenza like illness (General disorders and administration site conditions) | 2 | 0
Oedema peripheral (General disorders and administration site conditions) | 3 | 0
Pain (General disorders and administration site conditions) | 2 | 0
Pyrexia (General disorders and administration site conditions) | 18 | 0
Hepatic steatosis (Hepatobiliary disorders) | 2 | 0
COVID-19 (Infections and infestations) | 10 | 0
Influenza (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 9 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 0
Urinary tract infection (Infections and infestations) | 13 | 0
Alanine aminotransferase increased (Investigations) | 11 | 0
Amylase increased (Investigations) | 4 | 0
Aspartate aminotransferase increased (Investigations) | 17 | 0
Blood alkaline phosphatase increased (Investigations) | 4 | 0
Blood cholesterol increased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 8 | 0
Blood creatinine increased (Investigations) | 5 | 0
Blood glucose increased (Investigations) | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 4 | 0
Blood urea increased (Investigations) | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0
Lipase increased (Investigations) | 10 | 0
Lymphocyte count decreased (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 15 | 0
Platelet count decreased (Investigations) | 7 | 0
Urinary occult blood positive (Investigations) | 5 | 0
Weight decreased (Investigations) | 10 | 0
Weight increased (Investigations) | 6 | 0
White blood cell count decreased (Investigations) | 11 | 0
Decreased appetite (Metabolism and nutrition disorders) | 11 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 10 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 19 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 9 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 0
Dizziness (Nervous system disorders) | 5 | 0
Headache (Nervous system disorders) | 3 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Albuminuria (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 7 | 0
Proteinuria (Renal and urinary disorders) | 15 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 9 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 0
Hypertension (Vascular disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/77/NCT04452877/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT04452877/SAP_001.pdf